CLINICAL TRIAL: NCT07170384
Title: Evaluation of the Effect of the Mediterranean Diet on Disease Activity and Treatment Response in Patients With Axial Spondyloarthritis Receiving Biologic Therapy
Brief Title: Mediterranean Diet and Disease Activity in Axial Spondyloarthritis Receiving Biologic Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinem Kübra Beke (Other)
Responsible Party: Sponsor-Investigator, Sinem Kübra Beke, Associate Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS01
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Axial Spondyloarthritis (Ankylosing Spondylitis)
Keywords: Mediterranean Diet; Axial Spondyloarthritis; Ankylosing Spondylitis; Biologic Therapy; bDMARD
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized controlled trial using a parallel assignment model. Patients will be randomized into two groups: the intervention group receiving a Mediterranean diet program and the control group receiving standard care with general healthy eating advice
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. The outcomes assessor will be blinded to group allocation. Participants and care providers will be aware of the assigned intervention due to the nature of dietary modification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Group (Experimental): Participants will follow a structured Mediterranean diet program designed and supervised by a dietitian. Adherence will be reinforced through follow-up phone calls every 10 days. Assessments will be performed at baseline and after 3 months.
  Interventions: Behavioral: Mediterranean Diet
- Control Group (Standard Care) (Active Comparator): Participants will continue their standard medical treatment and will receive general healthy eating advice in addition to routine care. Assessments will be performed at baseline and after 3 months
  Interventions: Behavioral: Healthy Eating Advice

INTERVENTIONS:
Behavioral: Mediterranean Diet — "A structured Mediterranean diet program designed and supervised by a dietitian. The program emphasizes high consumption of olive oil, vegetables, fruits, legumes, whole grains, and fish; moderate intake of dairy and poultry; and low intake of red meat and processed foods. Adherence will be monitored through 10-day interval follow-up phone calls. Assessments will be conducted at baseline and 3 months
  Arms: Mediterranean Diet Group
Behavioral: Healthy Eating Advice — Participants will continue their standard medical treatment and will receive general healthy eating advice, as routinely recommended in clinical practice. No additional structured dietary program will be provided. Assessments will be performed at baseline and at 3 months.
  Arms: Control Group (Standard Care)

SUMMARY:
This study aims to evaluate the effect of the Mediterranean diet on disease activity, quality of life, inflammation, pain, and treatment response in patients with axial spondyloarthritis (ankylosing spondylitis) who are receiving stable biologic therapy. Axial spondyloarthritis is a chronic inflammatory disease that affects the spine and sacroiliac joints, often leading to pain, stiffness, and reduced quality of life. While biologic disease-modifying antirheumatic drugs (bDMARDs) are effective in reducing inflammation, lifestyle factors such as diet may also play an important role in disease outcomes.

In this randomized controlled trial, a total of 110 patients diagnosed with ankylosing spondylitis will be enrolled. Participants will be randomly assigned to either the Mediterranean diet group or the control group. The Mediterranean diet group will receive a structured diet program supervised by a dietitian, while the control group will continue their standard care with general healthy eating advice. Patients will be monitored for dietary adherence, and assessments will be conducted at baseline and after 3 months.

The primary outcome measure is the change in Ankylosing Spondylitis Disease Activity Score with C-reactive protein (ASDAS-CRP). Secondary outcomes include BASDAI, BASFI, BASMI, laboratory markers of inflammation, quality of life (SF-36), fatigue (FACIT-Fatigue), sleep quality (PSQI), anxiety and depression (HADS), medication adherence (MMAS-8), and Mediterranean diet adherence (PREDIMED). The study will provide valuable data on whether a Mediterranean diet can improve clinical outcomes and support the management of axial spondyloarthritis in patients receiving biologic therapy, potentially contributing to future lifestyle-based treatment strategies.

DETAILED DESCRIPTION:
Aim This study is designed to investigate the effects of the Mediterranean diet on disease activity, quality of life, inflammation levels, pain scores, and the frequency of biologic DMARD use in patients with ankylosing spondylitis (AS) receiving biologic disease-modifying antirheumatic drugs (bDMARDs).

Background Ankylosing spondylitis (AS) is a chronic inflammatory disease that causes early inflammation in the sacroiliac joints and, in later stages, also affects the axial skeleton. Structural and functional impairment, together with inflammatory back pain, lead to a marked reduction in quality of life. Genetic factors, intestinal microbiota, mechanical stress on the spine and peripheral joints, innate immunity, oxidative stress, lifestyle, and environmental influences are thought to play important roles in the pathogenesis of AS.

Both pharmacological and non-pharmacological strategies are used in the treatment of AS. The primary goal of treatment is to control symptoms and inflammation, prevent structural damage, and maximize long-term quality of life. However, there is limited evidence supporting the effectiveness of lifestyle modifications. Among environmental factors, diet is a modifiable component with the potential to reduce inflammation. Certain foods may trigger inflammatory processes, whereas nutrients such as antioxidants and omega-3 fatty acids may exert anti-inflammatory effects.

The Mediterranean diet (MD), with its anti-inflammatory and antioxidant potential, is considered a promising dietary model in chronic inflammatory conditions. This dietary pattern emphasizes high consumption of olive oil, unrefined carbohydrates, fresh and dried fruits, vegetables, and fish; low consumption of dairy products and red meat; and moderate consumption of red wine. In AS, such nutrients may reduce inflammation, alleviate pain, decrease structural damage, and potentially improve quality of life. No study has specifically compared the Mediterranean diet in AS patients receiving stable bDMARD therapy with a control group. This trial is intended to address this gap.

Hypothesis The investigators hypothesize that the Mediterranean diet will reduce disease activity, improve quality of life, and lower inflammation in patients with AS.

Study Design and Participants This study is designed as a prospective, single-blind, randomized controlled trial. The required sample size was calculated as 51 patients per group. Considering a 10% dropout rate, 55 patients will be included in each group, resulting in a total of 110 participants. Patients older than 18 years who meet the Assessment of SpondyloArthritis International Society (ASAS) classification criteria for AS will be eligible after providing written informed consent.

Inclusion Criteria

Diagnosis of AS according to ASAS criteria

Age ≥18 years

No dietary changes in the last 3 months

Stable treatment (NSAIDs or DMARDs) for the previous 4 months

Willingness to participate

Exclusion Criteria

Pregnancy or breastfeeding

Nutritional restrictions preventing adherence to the Mediterranean diet

Participation in another diet- or exercise-based intervention program within the last 6 months

History of other rheumatologic or neurological diseases

Patients meeting ASAS criteria for radiographic axial spondyloarthritis and aged over 18 years will be included after informed consent. Only those receiving biologic therapy for at least the previous 4 months with stable treatment will be enrolled.

Randomization and Blinding Participants will be randomized into intervention and control groups using stratified randomization according to age, body mass index, and disease activity (ASDAS-CRP). Randomization will be performed by an independent researcher using an online randomization system, with codes safeguarded to ensure allocation concealment. The outcome assessor will be blinded to group allocation.

Interventions

Control Group (Standard Care): Patients will continue routine medical treatment and will be advised to follow general healthy eating guidelines.

Mediterranean Diet Group: Patients will follow a structured Mediterranean diet program designed with a dietitian. Dietary adherence will be reinforced through telephone follow-ups every 10 days.

Assessments will be performed at baseline and at the end of the 3-month intervention.

Primary Outcome

Change in Ankylosing Spondylitis Disease Activity Score with C-reactive protein (ASDAS-CRP).

Secondary Outcomes

Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)

ASDAS using erythrocyte sedimentation rate (ASDAS-ESR)

Bath Ankylosing Spondylitis Functional Index (BASFI)

Bath Ankylosing Spondylitis Metrology Index (BASMI)

Hospital Anxiety and Depression Scale (HADS)

Quality of life (SF-36)

International Physical Activity Questionnaire (IPAQ)

Pittsburgh Sleep Quality Index (PSQI)

Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)

Health Assessment Questionnaire (HAQ)

Medication adherence (MMAS-8)

Mediterranean diet adherence (PREDIMED score)

Hand grip strength

Body composition analysis (InBody270 bioelectrical impedance analysis)

Power Analysis The required sample size was calculated using G*Power software with 80% power and a type I error of 0.05. A total of 55 participants per group was determined, accounting for a 10% dropout rate.

Statistical Analysis All analyses will be performed using SPSS software. The Shapiro-Wilk test will assess normality of data. Baseline characteristics will be compared using independent t-tests or Mann-Whitney U tests as appropriate. Repeated-measures ANOVA will be used for within- and between-group comparisons of primary and secondary outcomes at baseline and 3 months. Bonferroni correction will be applied for multiple comparisons. Categorical variables will be analyzed using Chi-square or Fisher's exact test. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.

Diagnosis of ankylosing spondylitis according to the Assessment of SpondyloArthritis International Society (ASAS) classification criteria.

No dietary changes within the past 3 months.

Stable treatment with NSAIDs or DMARDs for at least the previous 4 months.

Receiving biologic therapy (bDMARDs) with no changes in medication for the last 4 months.

Willingness and ability to provide written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding.

Nutritional restrictions preventing adherence to the Mediterranean diet (e.g., severe food allergies).

Participation in another diet- or exercise-based intervention program within the last 6 months.

Presence of another rheumatologic disease or history of neurological disorders.

Individuals younger than 18 years.

Contraindications to body composition analysis (e.g., cardiac pacemaker, pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score with C-reactive protein) | Baseline and 3 months
  ASDAS-CRP is a validated composite index for disease activity in ankylosing spondylitis. Disease activity states are classified as inactive (<1.3), low (<2.1), high (<3.5), and very high (>3.5). The primary outcome is the change in ASDAS-CRP score from baseline to 3 months.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline and 3 months
  BASDAI assesses fatigue, spinal pain, peripheral joint pain/swelling, localized tenderness, and morning stiffness (severity and duration) using six 10 cm visual analog scale (VAS) questions. Scores range from 0 (best) to 10 (worst).
th Ankylosing Spondylitis Functional Index (BASFI) | Baseline and 3 months
  BASFI evaluates functional ability through 10 daily activity questions scored on a 10 cm VAS. Higher scores indicate worse function.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Baseline and 3 months
  BASMI assesses spinal and hip mobility based on five measures: lateral lumbar flexion, tragus-to-wall distance, lumbar flexion, intermalleolar distance, and cervical rotation. Scores range from 0 (no limitation) to 10 (severe limitation).
Hospital Anxiety and Depression Scale (HADS) | Baseline and 3 months
  4-item questionnaire (7 anxiety, 7 depression). Scores >10 for anxiety (HADS-A) and >7 for depression (HADS-D) indicate possible mood disorder.
Quality of Life (Short Form-36, SF-36) | Baseline and 3 months
  SF-36 evaluates eight domains of health status (physical, role-physical, role-emotional, pain, general health, vitality, social, mental health). Scores 0-100; higher scores indicate better quality of life.
Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline and 3 months
  Self-reported questionnaire assessing sleep quality and disturbances over 1 month. Scores ≥5 indicate poor sleep quality.
Medication Adherence (Morisky Medication Adherence Scale, MMAS-8) | Baseline and 3 months
  8-item scale assessing adherence, categorized as low (<6), medium (6-7), or high (8).
Mediterranean Diet Adherence (PREDIMED Score) | Baseline and 3 months
  14-item questionnaire assessing adherence to the Mediterranean diet. Scores ≤5 = poor, 6-9 = moderate, ≥10 = good adherence.
Hand Grip Strength | Baseline and 3 months
  Measured with a calibrated Jamar hydraulic hand dynamometer for both dominant and non-dominant hands. The mean of three measurements will be recorded in kilograms.
Body Composition (InBody 270 Bioelectrical Impedance Analysis) | Baseline and 3 months
  Segmental skeletal muscle mass (arms, legs, trunk) will be assessed using multi-frequency bioelectrical impedance analysis (DSM-BIA).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Division of Rheumatology, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared due to patient privacy concerns and local data protection regulations. Only aggregate study results will be published in scientific journals and presented at conferences.

REFERENCES:
- [Result] Ometto F, Ortolan A, Farber D, Lorenzin M, Dellamaria G, Cozzi G, Favero M, Valentini R, Doria A, Ramonda R. Mediterranean diet in axial spondyloarthritis: an observational study in an Italian monocentric cohort. Arthritis Res Ther. 2021 Aug 20;23(1):219. doi: 10.1186/s13075-021-02600-0. PMID 34416917

DOCUMENTS (1):
  • Study Protocol (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT07170384/Prot_000.pdf